CLINICAL TRIAL: NCT04900922
Title: Changes in Shoulder Kinematics Following an Isokinetic Fatigue Protocol in Tennis Players
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Assistant professor, National Yang Ming Chiao Tung University
Other Study IDs: C109047
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Fatigue
Keywords: tennis player; shoulder kinematics; scapular kinematics; serving biomechanics; isokinetic dynamometer
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy tennis players: Participants in this group need to perform arm elevation in the scapular plane three times and successful flat tennis serve three times before and after a fatigue protocol. Surface electromyography on infraspinatus, pectoralis major, anterior deltoid ,and latissimus dorsi will be used to detect muscle activity related to fatigue.
  Interventions: Device: isokinetic dynamometer

INTERVENTIONS:
Device: isokinetic dynamometer — We will use an isokinetic dynamometer to conduct the concentric isokinetic fatigue protocol. The start position is shoulder abduction 90°, elbow flexion 90°and range of motion is set from 0 ° (internal rotation) to 90 ° (external rotation) under 120°/s. To calculate maximum torque of shoulder external and internal rotation, the subject will perform maximum isokinetic test 5 times before fatigue. Fatigue protocol include 10 sets, and each set include 32 repetitions with 30 seconds of rest between sets. The fatigue protocol will be stopped under three conditions: 1. the torque decreases 50% of maximum torque three times in one set or 2.rating of perceived exertion (RPE) abrove 15 and players can not perform the fatigue protocol or 3. finish the whole test.

SUMMARY:
A typical tennis match can take 1 to 5 hours. Tennis serve can be divided into eight stages and three phases. Injuries usually happen in the cocking stage and acceleration phase of the serve, where it requires large shoulder range of motion and proper scapular motion, including sufficient scapular upper rotation, external rotation, and posterior tilt to produce a powerful serve. Altered shoulder kinematics are associated with shoulder injuries in tennis players, including delayed shoulder horizontal adduction, and early external rotation. Due to the long duration and repetition of activity in a match, fatigue may happen and result in decreases in sensory input, passive range of motion, ball speed, and muscle strength. These changes may further lead to altered glenohumeral and scapular kinematics. However, previous studies mainly focused on the effects of fatigue on scapular kinematics in constrain movements and applied different fatigue protocols, which lead to inconsistent results. Tennis serve in cocking stage and the acceleration phase require high activation of shoulder external rotators and internal rotators, including infraspinatus, pectoralis major, subscapularis, latissimus dorsi and serratus anterior. However, to our knowledge, no study has investigated how fatigue of shoulder rotators influences shoulder kinematic as well as scapular kinematics during the late cocking stage and acceleration phase of tennis serve. Therefore, the investigators aim to investigate whether fatigue of shoulder rotator affects shoulder kinematics in healthy tennis players during the late cocking stage and acceleration phase of tennis serve.This is a single group, pretest-posttest measurement study. In a fatigue protocol, investigators use an isokinetic dynamometer to induce fatigue of shoulder rotators. Outcome measures will be tested before and after the fatigue protocol, including peak torque of shoulder rotators, humerothoracic kinematics, scapulothoracic kinematics, and median power frequency recorded by a surface electromyography. Peak torque of shoulder rotators will be measured with an isokinetic dynamometer. Surface electromyography will be used to measure peripheral muscle fatigue by maximum voluntary isometric contraction. Humerothoracic kinematics and scapulothoracic kinematics during a functional tennis serve and scaption will be collected with a motion capture system.

ELIGIBILITY:
Inclusion Criteria:

Healthy tennis players

1. Age ranges from 20-45 years old
2. Engaging in tennis for at least 1 year
3. Routine training 3 times a week
4. No history of cervical and/or shoulder injury in the past one year, or injury with VAS (visual analog pain scale) lower than 3 and without cervical-shoulder pain 7 days before testing
5. No operation on the shoulder, no shoulder subluxation, labral tear, and rotator cuff tear.
6. Neer's test, empty can test, and Hawkins Kennedy test are negative.

Exclusion Criteria:

1. History of cervical and/or shoulder injury in the past one year, or injury with VAS (visual analog pain scale) bigger than 3 and with cervical-shoulder pain 7 days before testing
2. Operation on the shoulder, history of shoulder subluxation, labral tear, and rotator cuff tear.
3. One of the three test results is positive: Neer's test, empty can test, and Hawkins Kennedy test.
4. Perform upper extremity resist training and tennis training 24 hours before testing.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All of the subjects are healthy during the test to avoid the risk of injury.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Serve sequence pattern | immediately after the intervention (fatigue protocol)
  Including the timing of shoulder horizontal adduction above 0 degree and the timing of shoulder external rotation above 90 degree during a tennis serve. Time would be normalized into 100 percentage and calculate the difference between shoulder horizontal adduction and external rotation described with percentage (%).
Scapular kinematics | immediately after the intervention (fatigue protocol)
  Including anterior/posterior tilt, upward/downward rotation, and internal/external rotation during arm elevation in scapular plane at 30°, 60°, 90°, and 120°, and during late cocking stage of tennis serve and at the end of acceleration phase of the serve. Scapulothoracic kinematics will be calculated and will be described with degree (°).
Shoulder kinematics | immediately after the intervention (fatigue protocol)
  Including shoulder external/internal rotation, horizontal adduction/abduction, elevation in the cocking stage of tennis serving and at the end of acceleration phase,will be calculated and will be described with degree (°).

SECONDARY OUTCOMES:
Median frequency | immediately after the intervention (fatigue protocol)
  The median frequency calculated from electromyographic data of infraspinatus, pectoralis major, anterior deltoid, and latissimus dorsi. The percentage change in median frequency will be calculated and will be described with percentage (%).
Shoulder internal and external rotation torque | immediately after the intervention (fatigue protocol)
  The first three and the last three of shoulder rotation torque will be recorded and be described with Newton metre (Nm).
Relative fatigue ratio | immediately after the intervention (fatigue protocol)
  Last three torque of shoulder external rotation and internal rotation will be divided by the first three torque of shoulder external rotation and internal rotation described with percentage (%).
ER/IR ratio | immediately after the intervention (fatigue protocol)
  The torque of shoulder external rotation divided by the torque of shoulder internal rotation and will be described with ratio before and after fatigue protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- Fu Jen catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided